CLINICAL TRIAL: NCT05124444
Title: TOlerance MOlecular and Genome-wide Studies With Renal Allograft Recipient Material
Acronym: TOMOGRAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: DESCARTES Working Group On Transplantation (Other)
Responsible Party: Principal Investigator, Annick Massart, Principal investigator, Université Libre de Bruxelles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015/379
Record Dates: First submitted 2021-11-01; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Sequence Analysis, RNA

STUDY DESIGN:
Intervention Model Description: 1. Exome-wide association study
  2. Transcriptomic analyses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (tolerant patients) (Experimental)
  Interventions: Genetic: High throughput DNA and RNA sequencing
- Controls (Experimental)
  Interventions: Genetic: High throughput DNA and RNA sequencing

INTERVENTIONS:
Genetic: High throughput DNA and RNA sequencing — High throughput DNA and RNA sequencing

SUMMARY:
TOMOGRAM is a European multicentric, prospective, experimental, controlled study that aims to increase our understanding of the causative mechanisms of operational tolerance in kidney transplantation through the achievement of several multimodal whole-genomic analysis in human biological samples.

ELIGIBILITY:
Inclusion Criteria:

* recipient of an allogenic renal allograft,
* have experienced (whatever ongoing or not) at least a whole year with blood creatinine <1.7 mg/dL and proteinuria </=1g/day or /g creatinine despite the COMPLETE discontinuation of immunosuppressive drugs,
* alternatively, have experienced (whatever ongoing or not) at least a whole year with stable blood creatinine (max 20% variation) and proteinuria above these criteria despite the COMPLETE discontinuation of immunosuppressive drugs

Exclusion Criteria:

* Past medical history of allogeneic bone-marrow transplantation / combined organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08-22 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Number of moderately to highly damaging exonic variants | Through study completion, an average of 2 year

REFERENCES:
- [Derived] Massart A, Danger R, Olsen C, Emond MJ, Viklicky O, Jacquemin V, Soblet J, Duerinckx S, Croes D, Perazzolo C, Hruba P, Daneels D, Caljon B, Sever MS, Pascual J, Miglinas M; Renal Tolerance Investigators; Pirson I, Ghisdal L, Smits G, Giral M, Abramowicz D, Abramowicz M, Brouard S. An exome-wide study of renal operational tolerance. Front Med (Lausanne). 2023 May 17;9:976248. doi: 10.3389/fmed.2022.976248. eCollection 2022. PMID 37265662